CLINICAL TRIAL: NCT04854408
Title: the Effect of Coronavac Vaccine (Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2 Vaccine) on Healthcare Workers' Menstrual Patterns
Brief Title: Evaluation of the Effect of Coronavac Vaccine (Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2 Vaccine) on Healthcare Workers' Menstrual Patterns
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Coronavacendometrium
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Vaccine Reaction; Coronavirus; Menstrual Problem; Endometrium
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Menstruation Disturbances | interventions — Health Personnel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: healthcare workers with the coronavac vaccine — Health workers who are vaccinated will fill in the 20-question survey electronically.

SUMMARY:
Coronavac, one of the vaccines developed within the scope of combating the COVID-19 pandemic that has surrounded the world for a year, started to be applied in the first healthcare workers in our country. In this important step taken to end the pandemic, information on vaccines is still limited. Most vaccines, including the Coronavac vaccine, are applied with approval for emergency use before phase 3 studies are fully completed. While investigating the effect of the vaccine on the virus, possible side effects should also be considered. In this context, it is not known whether the vaccine has an effect on the menstrual cycle, especially of women of reproductive age.

Our primary aim in our study is to evaluate the effect of the vaccine on the menstrual cycle and if the vaccine has any effect on the menstrual cycle, what kind of changes this effect causes.

DETAILED DESCRIPTION:
The survey contains 20 questions aimed at obtaining information about the menstrual cycles of health workers before and after vaccination. Demographic data of the participants are also taken.

ELIGIBILITY:
Inclusion Criteria:

* be positive for covid-19 (severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 )
* Having 1 or 2 doses of vaccine
* have menstruation
* Being a female health worker
* not using drugs that can affect menstruation

Exclusion Criteria:

* be negative for covid-19(severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 )
* have no menstruation
* Being a male health worker

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: It includes female healthcare workers between the ages of 8 and 45. For participation, 1 or 2 doses of vaccine should be administered and at least one menstrual period after the match.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Possible effects of Coronavac vaccine (severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 vaccine) on menstrual cycle | 40 days
  The change in the menstrual cycle of vaccinated healthcare workers after the first or the second dose is questioned with 20 questions. The content of the question consists of yes and no questions explaining the general epidemiological data of the patients and the amount of menstruation. These questions question the amount and change of menstruation before and after the vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided